CLINICAL TRIAL: NCT02236702
Title: Kappa Opioid Receptor Imaging in Depression (KOR Depression)
Status: Terminated | Type: Observational
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: S14-00643
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: Major Depressive Disorder; Anhedonia; Positron Emission Tomography (PET); Kappa Opioid Receptor (KOR)
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Asymptomatic control: Asymptomatic control
  Interventions: Other: Positron Emission Tomography (PET) imaging
- Mildly symptomatic with depressive symptoms: Mildly symptomatic with depressive symptoms
  Interventions: Other: Positron Emission Tomography (PET) imaging
- Moderately symptomatic with depressive symptoms: Moderately symptomatic with depressive symptoms
  Interventions: Other: Positron Emission Tomography (PET) imaging
- Severely symptomatic with depressive symptoms: Severely symptomatic with depressive symptoms
  Interventions: Other: Positron Emission Tomography (PET) imaging

INTERVENTIONS:
Other: Positron Emission Tomography (PET) imaging — Positron Emission Tomography (PET) imaging

SUMMARY:
The purpose of this study is to use positron emission tomography (PET) imaging to measure the activity of the kappa opioid receptor (KOR) in the brains of depressed and non-depressed individuals.

DETAILED DESCRIPTION:
The kappa opioid receptor (KOR) has been implicated in the etiology of fear, threat, and anhedonia in animal models of human depression psychopathology. Herein, we propose to study the KOR in vivo using positron emission tomography, and we will also measure the activity of the hypothalamic-pituitary-adrenal (HPA)-axis in all study participants. We propose to recruit up to N=50 medication-free individuals using a transdiagnostic approach, measure their KOR-selective radioligand [11C]LY2795050 volumes of distribution (VT), an equivalent of KOR availability using positron emission tomography (PET) and study the role of the KOR in mediating the quality and severity of the depressive phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for all subjects include a willingness to participate in a psychiatric evaluation, collection of behavioral ratings and neuroendocrine assessments, and imaging studies including 1 positron emission tomography (PET) scan and 1 mantic resonance imaging (MRI) scan.
2. We propose to use a transdiagnostic approach where participants will be stratified according to their symptom severity to have a full representation of different depressive severities and components of the depressive phenotype in the cohort. To ensure recruitment of participants from each level of this phenotype, we will employ a stratified sampling approach to recruit 12 participants who are asymptomatic (i.e., Montgomery-Asberg Depression Rating Scale (MADRS) score=0-6); 12 who are mildly symptomatic (i.e., MADRS score=7-19; 12 who are moderately symptomatic (i.e., MADRS sore=20-34); and 12 who are severely symptomatic (i.e., MADRS score>34).

Exclusion Criteria:

1. any major medical (including HIV due to possible neuropsychiatric affects; and asthma or heart disease which may limit the interpretation of the imaging results, for example due to changes in tracer delivery in hypertensive patients or significant weight change in prior 12 weeks prior to the study) and neurological illness or injury (i.e. head trauma with loss of consciousness);
2. any current or prior clinically significant substance use disorder (abuse and dependence within a year from imaging studies) as determined by Structured Clinical Interview for Diagnostic and Statistical Manual Disorders (SCID) interview;
3. acute or chronic suicidality as determined by the SCID interview;
4. presence of any legal or illegal psychoactive substances determined with urine toxicology, urine cotinine, carbon monoxide (CO) monitoring, and breathalyzer;
5. intelligence quotient (IQ) <70 based on past intelligence testing;
6. any metal in body that would pose a risk with MRI;
7. claustrophobia that would interfere with MRI or PET imaging;
8. pregnancy or nursing for women;
9. women with estrogen and/or progesterone levels outside the normal range, on birth control pills, peri- and post- menopausal women, and those with ovarectomies;
10. obesity as defined by a body mass index (BMI) of > 35;
11. use of psychoactive medications including regular use of benzodiazepines;
12. having an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participation in the study;
13. life-time history of use and abuse of opioids; and
14. presence of psychotic symptoms in patients with mood and anxiety disorders, schizophrenia or schizoaffective disorders; and
15. blood donation within 8 weeks prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are between the ages of 18-55, are medically healthy and not currently taking any medications to treat any medical illness, have been diagnosed with major depressive disorder (MDD) or will be as a result of this study, or are healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
[11C]LY2795050 volume of distribution (VT) values in specific brain regions of asymptomatic vs mildly symptomatic vs moderately symptomatic vs severely symptomatic individuals | one month
  To use the KOR radioligand [11C]LY2795050 and PET to examine the relation between KOR availability in the ventral striatum and amygdala, and the full dimensional spectrum of threat and loss symptomatology, and reward responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States